CLINICAL TRIAL: NCT05973552
Title: Assessment of Iron Absorption and Requirements During Pregnancy and Lactation in Kenyan Women
Brief Title: Iron Absorption and Requirements in Pregnancy and Lactation
Acronym: PILLAR_II
Status: Recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Columbia University (Other); Jomo Kenyatta University of Agriculture and Technology (Other); Msambweni County Referral Hospital (Unknown); ETH Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: PILLAR_II
Record Dates: First submitted 2023-07-18; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-06

CONDITIONS: Iron Requirements; Pregnancy; Lactation; Infancy; Iron Absorption
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- All participants: Women (n=250), are followed throughout their pregnancy. Mother-infant pairs are followed throughout the first 6-months postpartum. Women receive daily oral iron supplementation during pregnancy in accordance with local standards of care. Using the stable iron isotopes dilution methodology, concentration of the stable iron isotope tracer (57Fe) in circulation will be measured throughout pregnancy and up to 6 months postpartum in both, mother and infant.
  Interventions: Other: CO-rebreathing
- Randomly selected sub-group: To directly assess dietary iron absorption, in a randomly selected subset of women (n=35), oral and intravenous stable iron isotope tracers (54Fe, 58Fe) will be administered. Oral iron absorption and erythrocyte iron incorporation will be measured 14 days after tracer administration.
  Interventions: Other: CO-rebreathing; Other: Oral iron isotope administration (54Fe); Other: Intravenous iron isotope administration (58Fe)

INTERVENTIONS:
Other: CO-rebreathing — In the CO-rebreathing method, a dedicated apparatus is used for inhaling and rebreathing a very small bolus of CO through a spirometer for ~2 min, which is absorbed through the lungs and binds to Hb, and then the increase of HbCO content of blood is measured 8 min after the CO inhalation. The increase of COHb in blood samples can then be used to precisely calculate Hb mass and blood volume
Other: Oral iron isotope administration (54Fe) — Participants randomly assigned to the sub-group, will receive 54Fe with a test meal in the second and third trimester for assessment of dietary iron absorption
  Groups: Randomly selected sub-group
Other: Intravenous iron isotope administration (58Fe) — Participants randomly assigned to the sub-group, will receive intravenous 58Fe in the second and third trimester for assessment of erythrocyte iron incorporation
  Groups: Randomly selected sub-group

SUMMARY:
Iron requirements increase significantly during pregnancy. Current recommendations for iron intake in pregnant and lactating women (PLW) are mainly based on factorial estimates and extrapolated from non-PLW. High-quality quantitative data on iron requirements in PLW are lacking, particularly in Sub- Saharan Africa where anaemia and infections are common.

The primary objective of this study is to use the stable iron isotope technique to determine iron requirements and assess iron absorption and losses in PLW living in Kenya.

In this prospective observational study, we will enrol pregnant women in the first trimester (n = 250) from a previous study cohort (n=1000) who participated in an iron absorption study at least 12 months ago and received the stable iron (Fe) isotope 57Fe. This 57Fe has now distributed and equilibrated throughout the women's body iron. Once enrolled in the present study, following Kenyan guidelines, women will receive standard prenatal care, including routine daily iron and folate supplementation. We will collect venous blood samples in each trimester and at delivery, and during the first 6 months of lactation in the mothers and infants (heel prick samples). To directly assess dietary iron absorption, in a randomly selected subset of women (n=35), oral and intravenous stable iron isotope tracers (54Fe, 58Fe) will be administered in the 2nd and 3rd trimesters.

ELIGIBILITY:
Inclusion Criteria:

* Providing consent to the informed consent form
* Participation in a previous stable isotope absorption study and having received an oral dose of 15 mg 57Fe at least 12 months prior to the date of inclusion in the study
* Positive pregnancy test and gestational age <10 weeks based on history of last menstrual period
* Permanent residence in the study area, and not expected to leave the study site for more than 4 weeks over the following 16 months
* Assessment of good health by professional staff at Msambweni Hospital

Exclusion Criteria:

* Pre-pregnancy body mass index >30 kg/m2
* Blood transfusion or intravenous iron treatment within 4 months of study start
* Major chronic infectious disease (e.g., tuberculosis, HIV+, hepatitis)
* Major chronic non-infectious disease (e.g., Type 1 or 2 diabetes, cancer)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will recruit 250 pregnant women in the first trimester who previously participated in a stable iron isotope study (Clinical Trial ID: NCT05266703) and received 15 mg of the stable iron isotope 57Fe as an oral dose of ferrous sulphate at least 12 months before being enrolled in this trial.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-07-31 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Iron absorbed, lossed and gained in the first trimester | Change in 57Fe tracer abundance between gestational age 6, 10 and 15 weeks
  isotope dilution
Iron absorbed, lossed and gained in the second trimester | Change in 57Fe tracer abundance between gestational age 15, 20 and 25 weeks
  isotope dilution
Iron absorbed, lossed and gained in the third trimester | Change in 57Fe tracer abundance between gestational age 25, 30 and 35 weeks
  isotope dilution
Iron absorbed, lossed and gained throughout pregnancy | Change in 57Fe tracer abundance between gestational age 6, 10, 15, 20, 25, 30 and 35 weeks
  isotope dilution
Iron absorbed, lossed and gained in lactating women | Change in 57Fe tracer abundance between 6, 14 and 24 weeks postpartum
  isotope dilution
Iron absorbed, lossed and gained in infancy | Change in 57Fe tracer abundance between age 6, 14 and 24 weeks
  isotope dilution

SECONDARY OUTCOMES:
Fractional iron absorption (%) in the second trimester | gestational age 20 weeks
  shift in iron isotopic ratios
Fractional iron absorption (%) in the third trimester | gestational age 30 weeks
  shift in iron isotopic ratios
Erythrocyte iron incorporation (%) in the second trimester | gestational age 20 weeks
  shift in iron isotopic ratios
Erythrocyte iron incorporation (%) in the third trimester | gestational age 30 weeks
  shift in iron isotopic ratios
Hemoglobin concentration (g/dl) | gestational age 6 weeks
  Hb
Hemoglobin concentration (g/dl) | gestational age 10 weeks
  Hb
Hemoglobin concentration (g/dl) | gestational age 15 weeks
  Hb
Hemoglobin concentration (g/dl) | gestational age 20 weeks
  Hb
Hemoglobin concentration (g/dl) | gestational age 25 weeks
  Hb
Hemoglobin concentration (g/dl) | gestational age 30 weeks
  Hb
Hemoglobin concentration (g/dl) | gestational age 36 weeks
  Hb
Hemoglobin concentration (g/dl) | 6 weeks postpartum
  mother
Hemoglobin concentration (g/dl) | age 6 weeks
  infant
Hemoglobin concentration (g/dl) | 14 weeks postpartum
  mother
Hemoglobin concentration (g/dl) | age 14 weeks
  infant
Hemoglobin concentration (g/dl) | 24 weeks postpartum
  mother
Hemoglobin concentration (g/dl) | age 24 weeks
  infant
Mean corpuscular volume (fl) | gestational age 6 weeks
  MCV
Mean corpuscular volume (fl) | gestational age 10 weeks
  MCV
Mean corpuscular volume (fl) | gestational age 20 weeks
  MCV
Mean corpuscular volume (fl) | gestational age 30 weeks
  MCV
Mean corpuscular volume (fl) | 6 weeks postpartum
  mother
Mean corpuscular volume (fl) | age 6 weeks
  infant
Mean corpuscular volume (fl) | 14 weeks postpartum
  mother
Mean corpuscular volume (fl) | age 14 weeks
  infant
Mean corpuscular volume (fl) | 24 weeks postpartum
  mother
Mean corpuscular volume (fl) | age 24 weeks
  infant
Erythropoietin concentration (mU/ml) | gestational age 10 weeks
  EPO
Erythropoietin concentration (mU/ml) | gestational age 20 weeks
  EPO
Erythropoietin concentration (mU/ml) | gestational age 30 weeks
  EPO
Erythropoietin concentration (mU/ml) | 6 weeks postpartum
  EPO
Erythropoietin concentration (mU/ml) | 14 weeks postpartum
  EPO
Erythropoietin concentration (mU/ml) | 24 weeks postpartum
  EPO
Erythroferrone concentration (ng/ml) | gestational age 10 weeks
  ERFE
Erythroferrone concentration (ng/ml) | gestational age 20 weeks
  ERFE
Erythroferrone concentration (ng/ml) | gestational age 30 weeks
  ERFE
Erythroferrone concentration (ng/ml) | 6 weeks postpartum
  ERFE
Erythroferrone concentration (ng/ml) | 14 weeks postpartum
  ERFE
Erythroferrone concentration (ng/ml) | 24 weeks postpartum
  ERFE
Hepcidin concentration (ng/ml) | gestational age 10 weeks
  Hep
Hepcidin concentration (ng/ml) | gestational age 20 weeks
  Hep
Hepcidin concentration (ng/ml) | gestational age 30 weeks
  Hep
Hepcidin concentration (ng/ml) | 6 weeks postpartum
  Hep
Hepcidin concentration (ng/ml) | 14 weeks postpartum
  Hep
Hepcidin concentration (ng/ml) | 24 weeks postpartum
  Hep
Serum ferritin concentration (ug/l) | gestational age 10 weeks
  SF
Serum ferritin concentration (ug/l) | gestational age 20 weeks
  SF
Serum ferritin concentration (ug/l) | gestational age 30 weeks
  SF
Serum ferritin concentration (ug/l) | 6 weeks postpartum
  mother
Serum ferritin concentration (ug/l) | age 6 weeks
  infant
Serum ferritin concentration (ug/l) | 14 weeks postpartum
  mother
Serum ferritin concentration (ug/l) | age 14 weeks
  infant
Serum ferritin concentration (ug/l) | 24 weeks postpartum
  mother
Serum ferritin concentration (ug/l) | age 24 weeks
  infant
Soluble transferrin receptor concentration (ul/l) | gestational age 10 weeks
  sTfR
Soluble transferrin receptor concentration (ul/l) | gestational age 20 weeks
  sTfR
Soluble transferrin receptor concentration (ul/l) | gestational age 30 weeks
  sTfR
Soluble transferrin receptor concentration (ul/l) | 6 weeks postpartum
  mother
Soluble transferrin receptor concentration (ul/l) | age 6 weeks
  infant
Soluble transferrin receptor concentration (ul/l) | 14 weeks postpartum
  mother
Soluble transferrin receptor concentration (ul/l) | age 14 weeks
  infant
Soluble transferrin receptor concentration (ul/l) | 24 weeks postpartum
  mother
Soluble transferrin receptor concentration (ul/l) | age 24 weeks
  infant
C-reactive protein concentration (mg/l) | gestational age 10 weeks
  CRP
C-reactive protein concentration (mg/l) | gestational age 20 weeks
  CRP
C-reactive protein concentration (mg/l) | gestational age 30 weeks
  CRP
C-reactive protein concentration (mg/l) | 6 weeks postpartum
  mother
C-reactive protein concentration (mg/l) | age 6 weeks
  infant
C-reactive protein concentration (mg/l) | 14 weeks postpartum
  mother
C-reactive protein concentration (mg/l) | age 14 weeks
  infant
C-reactive protein concentration (mg/l) | 24 weeks postpartum
  mother
C-reactive protein concentration (mg/l) | age 24 weeks
  infant
alpha-glycoprotein concentration (mg/dl) | gestational age 10 weeks
  AGP
alpha-glycoprotein concentration (mg/dl) | gestational age 20 weeks
  AGP
alpha-glycoprotein concentration (mg/dl) | gestational age 30 weeks
  AGP
alpha-glycoprotein concentration (mg/dl) | 6 weeks postpartum
  mother
alpha-glycoprotein concentration (mg/dl) | age 6 weeks
  infant
alpha-glycoprotein concentration (mg/dl) | 14 weeks postpartum
  mother
alpha-glycoprotein concentration (mg/dl) | age 14 weeks
  infant
alpha-glycoprotein concentration (mg/dl) | 24 weeks postpartum
  mother
alpha-glycoprotein concentration (mg/dl) | age 24 weeks
  infant
Blood volume (l) | gestational age 10 weeks
Blood volume (l) | gestational age 20 weeks
  BV
Blood volume (l) | gestational age 30 weeks
  BV
Blood volume (l) | 6 weeks postpartum
  BV
Blood volume (l) | 14 weeks postpartum
  BV
Blood volume (l) | 24 weeks postpartum
  BV
Intestinal fatty acid binding protein | gestational age 10 weeks
  I-FABP
Intestinal fatty acid binding protein | gestational age 20 weeks
  I-FABP
Intestinal fatty acid binding protein | gestational age 30 weeks
  I-FABP
Retinol binding protein | gestational age 10 weeks
  RBP
Retinol binding protein | gestational age 20 weeks
  RBP
Retinol binding protein | gestational age 30 weeks
  RBP
soluble CD14 | gestational age 10 weeks
  sCD14
soluble CD14 | gestational age 20 weeks
  sCD14
soluble CD14 | gestational age 30 weeks
  sCD14
Insulin-like growth factor 1 | gestational age 10 weeks
  IGF-1
Insulin-like growth factor 1 | gestational age 20 weeks
  IGF-1
Insulin-like growth factor 1 | gestational age 30 weeks
  IGF-1
Fibroblast growth factor 21 | gestational age 10 weeks
  FGF21
Fibroblast growth factor 21 | gestational age 20 weeks
  FGF21
Fibroblast growth factor 21 | gestational age 30 weeks
  FGF21

CONTACTS AND LOCATIONS:
Locations (1):
- Msambweni Referral Hospital, Msambweni, Kenya

IPD SHARING:
Plan to Share IPD: No